CLINICAL TRIAL: NCT04401748
Title: A Randomized, Double-Blind, Phase 3 Study Evaluating the Safety and Efficacy of Venetoclax in Combination With Azacitidine in Patients Newly Diagnosed With Higher-Risk Myelodysplastic Syndrome (Higher-Risk MDS)
Brief Title: Study Of Venetoclax Tablet With Intravenous or Subcutaneous Azacitidine to Assess Change in Disease Activity In Adult Participants With Newly Diagnosed Higher-Risk Myelodysplastic Syndrome
Acronym: Verona
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-954; 2023-507153-16-00 (Other: EU CT)
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: MDS; Myelodysplastic Syndrome; Venetoclax; Azacitidine; AZA; Venclexta
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Venetoclax + Azacitidine (AZA) (Experimental): Participants will receive venetoclax once daily (QD) (Days 1-14) in combination with AZA QD (7 days of the first 9 days) of each 28 day cycle.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Arm 2: Placebo + Azacitidine (Active Comparator): Participants will receive placebo once daily (QD) (Days 1-14) in combination with AZA QD (7 days of the first 9 days) of each 28 day cycle.
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: Venetoclax — Tablet: Oral
  Other Names: ABT-199; GDC-0199; Venclexta
  Arms: Arm 1: Venetoclax + Azacitidine (AZA)
Drug: Azacitidine — Subcutaneous (SC) or Intravenous (IV) injection
  Other Names: AZA
Drug: Placebo — Tablet; Oral
  Arms: Arm 2: Placebo + Azacitidine

SUMMARY:
Myelodysplastic Syndrome (MDS) is a group of disorders that gradually affect the ability of a person's bone marrow (semi-liquid tissue present in many bones like backbones) to produce normal blood cells. Some people with MDS have a risk of the disease progressing to acute myeloid leukemia (AML), and a risk of death from the disease itself. Symptoms of MDS include fatigue, shortness of breath, unusual paleness due to anemia (low red blood cell count), easy or unusual bruising, and red spots just beneath the skin caused by bleeding. The purpose of this study is to see how safe and effective venetoclax and azacitidine (AZA) combination are when compared to AZA and a placebo (contains no medicine), in participants with newly diagnosed higher-risk MDS.

Venetoclax is an investigational drug being developed for the treatment of MDS. The study consists of two treatment arms - In one arm, participants will receive venetoclax and AZA. In another arm, participants will receive AZA and placebo. Adult participants with newly diagnosed higher-risk MDS will be enrolled. Around 500 participants will be enrolled in approximately 220 sites worldwide.

Participants in one arm will receive oral doses of venetoclax tablet and intravenous (infusion in the vein) or subcutaneous (given under the skin) AZA solution. Participants in another arm will receive oral doses of placebo tablet and intravenous or subcutaneous AZA solution.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood and bone marrow tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of Myelodysplastic Syndrome (MDS) according to the 2016 World Health Organization (WHO) classification wtih presence of < 20% bone marrow blasts per marrow biopsy/aspirate at screening.
* Participants must meet the following disease activity criteria:

  * Overall Revised International Prognostic Scoring System (IPSS-R) score > 3 (intermediate, high or very high).
  * Eastern Cooperative Oncology Group (ECOG) performance status of <= 2.
  * Hematopoietic stem cell transplant (HSCT) eligible with no pre-arranged HSCT at the time of Study Day 1, or HSCT ineligible without plan for HSCT at the time of Study Day 1.

Exclusion Criteria:

* Prior therapy for MDS with any hypomethylating agent, chemotherapy, or allogenic stem cell transplantation.
* Prior diagnosis of therapy-related MDS (t-MDS), MDS evolving from a pre-existing myeloproliferative neoplasm (MPN), MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up To 5 Years
  OS is defined as the number of days from the date of randomization to the date of death of any cause, or last known date to be alive.

SECONDARY OUTCOMES:
Modified Overall Response (mOR) | Up To 5 Years
  mOR [complete remission (CR) + marrow complete remission (mCR) + partial response (PR)] is defined as achieving a CR, mCR, or PR at any time point during the study per the modified International Working Group (IWG) 2006 criteria for myelodysplastic syndrome (MDS).
Percentage of Participants Achieving Overall Hematological Improvement (HI) | Up to 5 Years
  Overall HI is defined as achieving the response of HI-platelet or HI-neutrophil, or HI-erythroid at any time point during the study prior to post-treatment therapy per the modified IWG 2006 criteria for MDS.
Complete Remission (CR) | Up To 36 Months
  CR is defined as achieving a complete remission at any time point during the study per the modified International Working Group (IWG) 2006 criteria for myelodysplastic syndrome (MDS).
Percentage of Participants Achieving Transfusion Independence (TI) Who are Transfusion Dependent at Baseline | Up To 5 Years
  TI is when the participants who were transfusion dependent on red blood cell (RBC) and/or Platelet at baseline achieve transfusion independence post baseline. TI is a period of at least 56 days with no transfusion after the date of the first dose of study drug to the last dose of study drug + 30 days, or 1 day before the date of progressive disease/ relapse from CR or PR per the modified IWG 2006 criteria for MDS, or 1 day before the initiation of post-treatment therapy or 1 day before death, whichever is earliest.
Time to Deterioration in Physical Functioning as Measured by Physical Functioning Domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scale | Up To 5 Years
  Time to deterioration in physical functioning, as measured by the EORTC QLQ-C30 physical functioning score is defined as the time from the date of randomization to the date of death of any cause, or the first time worsening of score from baseline >= a pre-specified threshold. Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue Short Form (SF) 7a Scale Score | Up To 5 Years
  Fatigue will be assessed using the PROMIS Fatigue SF 7a Global Fatigue Score. PROMIS Fatigue SF 7a is a 7-item questionnaire that assesses the impact and experience of fatigue over the past 7 days. Participants rate items on a 5-point scale, with 1 as "never" an 5 as "always".
Overall Response (OR) | Up To 5 Years
  OR [complete remission (CR) + partial response (PR)] is defined as achieving a CR or PR at any time point during the study per the modified IWG 2006 criteria for MDS.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (220):
- United States (58):
  - Duplicate_Providence Medical Foundation /ID# 222633, Fullerton, California
  - University of California, Los Angeles /ID# 221760, Los Angeles, California
  - Torrance Memorial Physician Network Cancer Care /ID# 222702, Torrance, California
  - PIH Health Whittier Hospital /ID# 222647, Whittier, California
  - Rocky Mountain Cancer Centers - Boulder /ID# 223723, Boulder, Colorado
  - Yale University School of Medicine /ID# 222764, New Haven, Connecticut
  - Helen F. Graham Cancer Center & Research Institute /ID# 223731, Newark, Delaware
  - Florida Cancer Specialists - Fort Myers /ID# 221319, Fort Myers, Florida
  - Memorial Healthcare System /ID# 222703, Hollywood, Florida
  - Florida Cancer Specialists - North /ID# 221318, St. Petersburg, Florida
  - Florida Cancer Specialists - Panhandle /ID# 221315, Tallahassee, Florida
  - Florida Cancer Specialists - East /ID# 221317, West Palm Beach, Florida
  - St. Luke's Mountain State Tumor Institute /ID# 220838, Boise, Idaho
  - Northwestern University Feinberg School of Medicine /ID# 220843, Chicago, Illinois
  - Duplicate_Rush University Medical Center /ID# 221007, Chicago, Illinois
  - Ingalls Memorial Hosp /ID# 220844, Harvey, Illinois
  - Illinois Cancer Care, PC /ID# 220840, Peoria, Illinois
  - Duplicate_Parkview Cancer Institute /ID# 223620, Fort Wayne, Indiana
  - Cancer Center of Kansas /ID# 222648, Wichita, Kansas
  - Hematology/Oncology Clinic /ID# 224257, Baton Rouge, Louisiana
  - Pontchartrain Cancer Center - Covington /ID# 221005, Covington, Louisiana
  - Maryland Oncology Hematology /ID# 223776, Columbia, Maryland
  - Massachusetts General Hospital /ID# 225068, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 225069, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 219162, Boston, Massachusetts
  - VA Ann Arbor Healthcare System /ID# 221365, Ann Arbor, Michigan
  - Cancer & Hematology Centers /ID# 220848, Grand Rapids, Michigan
  - Metro Minnesota Community Oncology Research Consortium (MMCORC) /ID# 221321, Saint Louis Park, Minnesota
  - MidAmerica Division, Inc. /ID# 221895, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada - Horizon Ridge /ID# 222635, Henderson, Nevada
  - Titan Health Partners LLC, d/b/a Astera Cancer Care /ID# 221003, East Brunswick, New Jersey
  - The Valley Hospital /ID# 232337, Paramus, New Jersey
  - New York Oncology Hematology - Albany Cancer Center /ID# 223778, Albany, New York
  - University at Buffalo /ID# 221206, Buffalo, New York
  - Weill Cornell Medical College /ID# 222898, New York, New York
  - Stony Brook University Hospital /ID# 224450, Stony Brook, New York
  - Novant Health Presbyterian Medical Center /ID# 222561, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center /ID# 221004, Winston-Salem, North Carolina
  - Oncology Hematology Care, Inc. /ID# 223724, Cincinnati, Ohio
  - Bend Memorial Clinic /ID# 220999, Bend, Oregon
  - Willamette Valley Cancer Institute and Research Center /ID# 223733, Eugene, Oregon
  - UPMC Hillman Cancer Ctr /ID# 223201, Pittsburgh, Pennsylvania
  - Avera Cancer Institute /ID# 243461, Sioux Falls, South Dakota
  - Tennessee Oncology - Chattanooga / McCallie /ID# 221311, Chattanooga, Tennessee
  - Tennessee Oncology-Nashville Centennial /ID# 220854, Nashville, Tennessee
  - Texas Oncology - Austin Midtown /ID# 223729, Austin, Texas
  - Duplicate_Texas Oncology - Medical City Dallas /ID# 223725, Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 223727, Dallas, Texas
  - Texas Oncology - Forth Worth /ID# 223777, Fort Worth, Texas
  - MD Anderson Cancer Center at Texas Medical Center /ID# 219163, Houston, Texas
  - Texas Oncology - San Antonio Medical Center - Research Drive /ID# 223728, San Antonio, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 221332, Temple, Texas
  - Texas Oncology - Northeast Texas /ID# 223734, Tyler, Texas
  - Utah Cancer Specialists Salt Lake Clinic /ID# 219160, Salt Lake City, Utah
  - Virginia Cancer Specialists - Gainesville /ID# 223726, Gainesville, Virginia
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 221590, Richmond, Virginia
  - Virginia Cancer Institute at Reynolds Crossing /ID# 221002, Richmond, Virginia
  - VA Puget Sound Health Care System /ID# 221358, Seattle, Washington
- Australia (7):
  - Duplicate_Blacktown Hospital /ID# 234079, Blacktown, New South Wales
  - St George Hospital /ID# 221810, Kogarah, New South Wales
  - Port Macquarie Base Hospital /ID# 234078, Port Macquarie, New South Wales
  - Gold coast University Hospital /ID# 222606, Southport, Queensland
  - Royal Adelaide Hospital /ID# 221805, Adelaide, South Australia
  - St Vincent's Hospital Melbourne /ID# 221809, Fitzroy Melbourne, Victoria
  - Austin Health /ID# 221807, Heidelberg, Victoria
- Austria (5):
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 221387, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 221386, Wels, Upper Austria
  - Medizinische Universitaet Wien /ID# 221446, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 221092, Salzburg
  - Hanusch Krankenhaus /ID# 221093, Vienna
- Belgium (7):
  - ZAS Middelheim /ID# 218907, Antwerp, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 219066, Brussels, Brussels Capital
  - Hospital La Louviere Site Jolimont - Helora /ID# 218921, La Louvière, Hainaut
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 219064, Yvoir, Namur
  - UZ Gent /ID# 218767, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 218905, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge /ID# 218212, Bruges, West-Vlaanderen
- Brazil (5):
  - Hospital Universitario Walter Cantidio /ID# 223434, Fortaleza, Ceará
  - Hospital Erasto Gaertner /ID# 221341, Curitiba, Puerto Rico
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein /ID# 221370, São Paulo, São Paulo
  - Hospital Universitário Pedro Ernesto /ID# 223080, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 221339, São Paulo
- Canada (6):
  - BC Cancer - Surrey /ID# 219098, Surrey, British Columbia
  - Ottawa Hospital Research Institute /ID# 219105, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre /ID# 219103, Toronto, Ontario
  - McGill University Health Centre - Glen Site /ID# 222519, Montreal, Quebec
  - CIUSSS du Nord-de-l'ile-de-Montréal_Hopital du Sacré-Coeur de Montréal /ID# 218973, Montreal, Quebec
  - CHUQ- Hôpital de l'Enfant-Jesus /ID# 221200, Québec, Quebec
- China (23):
  - Peking University International Hospital /ID# 222987, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital /ID# 225980, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital /ID# 221442, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University /ID# 222071, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 224566, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 222919, Shijiazhuang, Hebei
  - People's Hospital of Henan Province /ID# 225790, Zhengzhou, Henan
  - Henan Cancer Hospital /ID# 221447, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 221475, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 221474, Wuhan, Hubei
  - Zhongda Hospital Southeast University /ID# 221849, Nanjing, Jiangsu
  - Jiangsu Province Hospital /ID# 221342, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 221640, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 225983, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University /ID# 222945, Shenyang, Liaoning
  - Shaanxi Provincial People'S Hospital /ID# 225728, Xi'an, Shaanxi
  - Shanghai Sixth People's Hospital /ID# 221546, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 221601, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 221567, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital /ID# 226810, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 221494, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 225982, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine /ID# 225918, Yiwu, Zhejiang
- Czechia (6):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 221351, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 221163, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 219143, Ostrava, Ostrava-mesto
  - Fakultní Nemocnice Plzeň-Lochotín /ID# 221162, Pilsen, Plzen-jih
  - Všeobecná Fakultní Nemocnice v Praze /ID# 221229, Prague, Praha 17
  - Ustav hematologie a krevni transfuze /ID# 221350, Prague
- France (9):
  - Chu de Nice-Hopital L'Archet Ii /Id# 220992, Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire de Bordeaux /ID# 220989, Pessac, Gironde
  - CHU Grenoble - Hopital Michallon /ID# 220988, La Tronche, Isere
  - CHRU Lille - Hopital Claude Huriez /ID# 220991, Lille, Nord
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 222074, Nantes, Pays de la Loire Region
  - Hopital de la Conception /ID# 224882, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Henri Becquerel /ID# 220986, Rouen, Seine-Maritime
  - CH Henri Duffaut /ID# 225185, Avignon, Vaucluse
  - Hôpital Saint-Louis /ID# 222075, Paris
- Germany (8):
  - Universitatsklinikum Mannheim /ID# 221172, Mannheim, Baden-Wurttemberg
  - Stauferklinikum Schwaebisch Gmuend /ID# 224917, Mutlangen, Baden-Wurttemberg
  - Klinikum rechts der Isar /ID# 221170, Munich, Bavaria
  - Medizinische Hochschule Hannover /ID# 221173, Hanover, Lower Saxony
  - Universitaetsklinikum Koeln /ID# 234219, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf /ID# 221169, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 221168, Leipzig, Saxony
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 221189, Berlin
- Hungary (5):
  - Fejér Vármegyei Szent György Egyetemi Oktató Kórház /ID# 222953, Székesfehérvár, Fejér
  - Duplicate_Debreceni Egyetem Klinikai Kozpont /ID# 221702, Debrecen, Hajdú-Bihar
  - Duplicate_Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 221703, Kaposvár, Somogy County
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 221704, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Szegedi Tudományegyetem /ID# 221705, Szeged
- Israel (6):
  - Shaare Zedek Medical Center /ID# 233181, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 222006, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 221110, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 221896, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 221083, Haifa
  - Rabin Medical Center /ID# 221184, Petah Tikva
- Italy (5):
  - IRCCS Istituto Clinico Humanitas /ID# 220815, Rozzano, Lombardy
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli /ID# 220816, Naples, Napoli
  - Duplicate_Azienda Ospedaliero-Universitaria Sant'Andrea /ID# 220819, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 220810, Bologna
  - Grande Ospedale Metropolitano Bianchi - Melacrino - Morelli P.O. Riuniti /ID# 220818, Reggio Calabria
- Japan (16):
  - Nagoya University Hospital /ID# 221566, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 221568, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 223473, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 222015, Fukushima, Fukushima
  - Chugoku Central Hospital /ID# 222955, Fukuyama, Hiroshima
  - Sapporo Hokuyu Hospital /ID# 222133, Sapporo, Hokkaido
  - Aiiku Hospital /ID# 222351, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 221977, Kobe, Hyōgo
  - NHO Mito Medical Center /ID# 222278, Higashiibaraki-gun, Ibaraki
  - Tohoku University Hospital /ID# 221976, Sendai, Miyagi
  - Okayama Medical Center /ID# 222310, Okayama, Okayama-ken
  - Kindai University Hospital /ID# 222284, Osakasayama-shi, Osaka
  - Saitama Medical Center /ID# 222016, Kawagoe, Saitama
  - NTT Medical Center Tokyo /ID# 222365, Shinagawa-ku, Tokyo
  - Yamagata University Hospital /ID# 221574, Yamagata, Yamagata
  - Nagasaki University Hospital /ID# 222241, Nagasaki
- Netherlands (5):
  - Maastricht Universitair Medisch Centrum /ID# 221630, Maastricht, Limburg
  - Maxima Medisch Centrum /ID# 223010, Eindhoven, North Brabant
  - Medisch Spectrum Twente /ID# 223012, Enschede, Overijssel
  - Isala /ID# 223011, Zwolle, Overijssel
  - Erasmus Medisch Centrum /ID# 218937, Rotterdam, South Holland
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela /ID# 233321, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie /ID# 221667, Lublin, Lublin Voivodeship
  - Lux Med Onkologia - Szpital Szamocka /Id# 222203, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by Pratia /ID# 221354, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne /ID# 222069, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice /ID# 224728, Katowice
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopern /ID# 221784, Lodz, Łódź Voivodeship
- Puerto Rico (2):
  - Pan American Center for Oncology Trials, LLC /ID# 221010, Rio Piedras
  - VA Caribbean Healthcare System /ID# 221012, San Juan
- Russia (6):
  - Kaluga Regional Clinical Hospital /ID# 221211, Kaluga, Kaluga Oblast
  - Republican hospital named after V.A. Baranov /ID# 221214, Petrozavodsk, Murmansk Oblast
  - Clinic UZI 4D /ID# 221215, Pyatigorsk, Stavropol Kray
  - Hospital n.a. V.V. Veresaev /ID# 225435, Moscow
  - MMCC Kommunarka /ID# 221213, Moscow
  - Almazov National Medical Research Centre /ID# 221449, Saint Petersburg
- South Korea (6):
  - Duplicate_Pusan National University Hospital /ID# 232353, Busan, Busan Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 221695, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 221226, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 221227, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 221224, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 233171, Seoul
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol /ID# 221274, Badalona, Barcelona
  - Hospital Universitario Reina Sofia /ID# 221273, Córdoba, Cordoba
  - Hospital Universitario Quironsalud Madrid /ID# 221275, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Vall d'Hebron /ID# 221323, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 221271, Madrid
  - Hospital Universitario 12 de Octubre /ID# 221272, Madrid
  - Hospital Universitario de Salamanca /ID# 221297, Salamanca
  - Hospital Universitario Virgen del Rocio /ID# 221276, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 221270, Valencia
- Taiwan (4):
  - Duplicate_Kaohsiung Chang Gung Memorial Hospital /ID# 223573, Kaohsiung City, Kaohsiung
  - China Medical University Hospital /ID# 218987, Taichung
  - National Cheng Kung University Hospital /ID# 218989, Tainan
  - Chi-Mei Medical Center /ID# 218991, Tainan
- Turkey (Türkiye) (6):
  - Duplicate_Erciyes University Medical Fac /ID# 222090, Melikgazi, Kayseri
  - Hacettepe University Faculty of Medicine /ID# 222094, Ankara
  - Ankara City Hospital /ID# 222093, Ankara
  - Akdeniz Universitesi Tip Fakul /ID# 222095, Antalya
  - Ondokuz mayis University Facul /ID# 222091, Samsun
  - Acibadem Maslak Hastanesi /ID# 222072, Tuzla
- United Kingdom (9):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 222514, Plymouth, Devon
  - University Hospitals Dorset NHS Foundation Trust /ID# 221237, Poole, Dorset
  - University College London Hospital /ID# 221240, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust /ID# 221231, Oxford, Oxfordshire
  - Cardiff & Vale University Health Board /ID# 221236, Cardiff, Wales
  - NHS Grampian /ID# 222509, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust /ID# 221233, Birmingham
  - University Hospitals Bristol /ID# 222510, Bristol
  - The Royal Marsden NHS Foundation Trust /ID# 221232, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Stahl M, DeZern AE. Is there a path forward for immunotherapy in patients with myelodysplastic syndromes? Lancet Haematol. 2024 Jan;11(1):e5-e7. doi: 10.1016/S2352-3026(23)00343-5. Epub 2023 Dec 5. No abstract available. PMID 38065202
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com